CLINICAL TRIAL: NCT06796400
Title: Effects of Theraband Versus General Exercises on Scapular Dyskinesia in Male Cricketers.
Brief Title: Effects of TBE VS GE on Scapular Dyskinesia in Male Cricketers.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RiphahIU/ m66icc nadia ishtiaq
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Scapular Dyskinesis
Keywords: Pain Scapular dyskinesia Strength Theraband exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General exercises (Active Comparator): Resistance based exercises with load for muscles strengthing.
  Interventions: Other: General exercises
- Theraband exercises (Experimental): Rubber based resistance exercises which target the specific muscles for strength.
  Interventions: Other: Theraband exerises

INTERVENTIONS:
Other: General exercises — 4 general exercises were done by control group with 10 repetitions and 3 sets, 6 times per week, up to 8 weeks.These exercises are for lower trapzius and serratus anterior mucles strengthing.
  Arms: General exercises
Other: Theraband exerises — 5 Thera-band exercises were completed by experimental group with 3 sets and 10 repetitions, 6 times per week, up to 8 weeks. These exercises are for lower trapzius and serratus anterior mucles strengthing.
  Arms: Theraband exercises

SUMMARY:
We wanted to find the effectiveness between the theraband and general exercises on scapular dyskinesis in male cricket players.

DETAILED DESCRIPTION:
Cricket game is considered a non-contact low-injury risk sport associated to other sports, chronic and acute traumatic injuries are the two common types of injury mechanisms. Theraband exercises are those exercises which are considered as a safe tool which increases the functional ability and muscle strength. Scapular dyskinesis (which is called as sick scapula) as commonly defined as an alteration or deviation in the resting position or during movable position of the scapula during shoulder joint motions. A study reported that Theraband exercises increase the function of the muscles. These muscles participate to the strength of the shoulder girdle, stability and mobility. Theraband exercises are considered to be able increase the proprioception and balance. The prevalence of scapular dyskinesia (74.6%) dominant side scapula turns medially, inferiorly, and also tilts anteriorly as relate to non-dominant side shoulder blade.Scapular dyskinesia has been more determined in healthy individuals but statics has also mentioned that scapular dyskinesia a greater prevalence in overhead (61%) than non-overhead sportspersons (33%). Maximum cricket players complain that they feel discomfort in the scapular region. Because occasionally the scapular dyskinesia causes the discomfort in scapula region and it is due to the muscles weakness of the scapula. It is mostly occur in overhead athletes because of the constant repetitions of the shoulder movement over the head. For intervention purpose in scapular dyskinesia, cricket players maximum concentrate on general exercises instead of theraband exercises because they don't aware about the effectiveness of theraband exercises in this condition and theraband exercises involve using resistance bands of varying strengths to perform specific movements targeting the muscles around the scapula. These exercises could help improve the muscle strength, endurance, and control, which will be essential for stabilizing the scapula and improving its movement patterns while general exercises improve the overall functional movement patterns, which may indirectly benefit scapular dyskinesia by strengthening surrounding muscles and improving overall shoulder mechanics. Despite up to my searched no study has been found about it so this study is designed to find the effectiveness of thera-band exercises on scapular dyskinesia in male cricketers.

ELIGIBILITY:
Inclusion Criteria:

* • Scapular dyskinesia type I

  * Only male cricketers.
  * Age from 18 to 30 years old.
  * Training at least 4 times per week and 10 hours weekly training.
  * Male cricket players playing since last one year.

Exclusion Criteria:

* • The history of scapular fracture repair surgery and neck surgery during previous 12 months.

  * The players that are out of practice from 5 weeks.
  * Traumatic history of cervical region and scapula.
  * Serious pathologies regarding shoulder, cervical and scapula.
  * Female cricketers

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male gender
Enrollment: 52 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-09-03 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Hand-held dynamometer | 8 week
  Handheld Dynamometry (HHD) is a procedure utilized to judge muscle strength. This version of a dynamometer is set up or held by the physical therapist to originate an objective measurement of force. The Scapular protraction test is usually used to measure the strength of the serratus anterior while Prone Scapular Retraction test is utilized to evaluate the strength of lower trapezius muscle then utilized a dynamometer to measure the force applied by the participant. A perfect reading on the dynamometer, with small asymmetry between sides, pretends normal serratus anterior function otherwise it will be abnormal.

SECONDARY OUTCOMES:
Numeric pain rating scale | 8 week
  The Numeric Pain Rating Scale, which is utilized in medical settings, permits persons to rate their pain on a scale from 0 to 10, with 0 representing that there is no pain and 10 showing the worst possible pain. The pain severity is evaluated by this scale

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Ishtiaq, MS, Principal Investigator — nadia.ishtiaq@riphah.edu.pk
Locations (1):
- JI youth cricket academy, peshawar, Peshawar, Khyber Pkhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No